CLINICAL TRIAL: NCT03919578
Title: Protectivity and Safety Following Recombinant Hepatitis B Vaccine With Different Source of Hepatitis B Bulk Compared to Hepatitis B (Bio Farma) Vaccine in Indonesian Population
Brief Title: Protectivity and Safety Following Recombinant Hepatitis B Vaccine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Hep B 0218
Record Dates: First submitted 2019-04-11; First posted 2019-04-18 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Immunogenicity
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Intervention Model Description: Experimental, randomized, double blind, four arm parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product was masking with control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hep B Batch 1 (Experimental): 1 dose of 1 mL Hepatitis B Batch 1
  Interventions: Biological: Recombinant Hepatitis B vaccine
- Hep B Batch 2 (Experimental): 1 dose of 1 mL Hepatitis B Batch 2
  Interventions: Biological: Recombinant Hepatitis B vaccine
- Hep B Batch 3 (Experimental): 1 dose of 1 mL Hepatitis B Batch 3
  Interventions: Biological: Recombinant Hepatitis B vaccine
- Hep B (Bio Farma) (Active Comparator): 1 dose of 1 mL Hepatitis B (Bio Farma)
  Interventions: Biological: Recombinant Hepatitis B (Bio Farma)

INTERVENTIONS:
Biological: Recombinant Hepatitis B vaccine — Recombinant Hepatitis B vaccine is an inactivated HbsAg produced in yeast cells (Hansenula polymorpha) using recombinant DNA technology. It is a whitish liquid produced by culture genetically engineered yeast cell which carry the relevant gene of the HbsAg. The inactivated HbsAg (bulk) is imported from Serum Institute of India and then formulated and filled at Bio Farma.
  Arms: Hep B Batch 1; Hep B Batch 2; Hep B Batch 3
Biological: Recombinant Hepatitis B (Bio Farma) — Recombinant Hepatitis B vaccine is an inactivated HbsAg produced in yeast cells (Hansenula polymorpha) using recombinant DNA technology. It is a whitish liquid produced by culture genetically engineered yeast cell which carry the relevant gene of the HbsAg. The inactivated HbsAg (bulk) is imported from The Janssen Vaccine Corp and then formulated and filled at Bio Farma.
  Arms: Hep B (Bio Farma)

SUMMARY:
Protectivity and Safety Following Recombinant Hepatitis B Vaccine with different source of Hepatitis B bulk compared to Hepatitis B (Bio Farma) vaccine in Indonesian Population

DETAILED DESCRIPTION:
Protectivity and Safety Following Recombinant Hepatitis B Vaccine with different source of Hepatitis B bulk compared to Hepatitis B (Bio Farma) vaccine in Indonesian Population.

Experimental, randomized, double blind, four arm parallel group study, lot to lot consistency study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individu as determined by clinical judgment, including a medical history and physical exam which confirms the absence of a current or past disease state considered significant by the investigator.
2. Subjects/parents/guardian(s) have been informed properly regarding the study and signed the informed consent form/ informed assent form.
3. Subject/parents/guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. Subjects with known history of Hepatitis B contained vaccination in the last 10 years
3. Evolving severe illness and/or chronic disease and fever (axillary temperature more than37.5oC) within the 48 hours preceding enrollment.
4. Known history of allergy to any component of the vaccines (based on anamnesis)
5. HBsAg positive
6. Known history of immunodeficiency disorder (HIV infection, leukemia, lymphoma, or malignancy).
7. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
8. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or corticosteroid therapy and other immunosuppresant.
9. Pregnancy & Lactation (Adult)
10. Subject already immunized with any vaccine within 4 weeks prior and expects to receive other vaccines within 4 weeks following immunization.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 536 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with increasing antibody titer >= 4 times | 28 days after the last dose immunization
  Percentage of subjects with increasing antibody titer >= 4 times: in all subjects; comparison between investigational product and control and between each lot number of Recombinant Hepatitis B

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) | 28 days after the last dose immunization
  GMT in all subjects; comparison of GMT between investigational products and control and comparison of GMT between each lot number of Recombinant Hepatitis B
Percentage of subjects with transition of seronegative to seropositive | 28 days after the last dose immunization
  Percentage of subjects with transition of seronegative to seropositive: in all subjects; Subjets which get investigational products and control and each lot number of Recombinant Hepatitis B
Percentage of subjects with at least one immediate reaction | 30 minutes after each vaccination
  Immediate reaction (local reaction or systemic event)
Percentage of subjects with at least one of these adverse events | within 72 hours, between 72 hours to 28 days after vaccination
  At least one of these adverse events, expected or not
Serious adverse event after vaccination | 28 days after the last dose immunization
  Serious adverse event occurring from inclusion until 28 days after vaccination.
Comparison adverse events between Investigational Products (Hepatitis B) and Control | 28 days after each dose
  Adverse events occuring until 28 days after vaccination
Comparison of adverse events between each lot number of Recombinant Hepatitis B vaccine | 28 days after each dose
  Adverse events occuring until 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yetty M Nency, MD, Principal Investigator — Universitas Diponegoro
Locations (1):
- RSND, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No